CLINICAL TRIAL: NCT06591234
Title: A Multicenter Study on the Reliability of Four Ultrasound Measures : the Antero-posterior Diameter , the End-exipratory Area , the Aspect Ratio and the Collapsibility Index of Internal Jugular Vein Evaluated on Images Recorded From Patients Admitted to Four Medicine Departments
Brief Title: Reliability of Internal Jugular Ultrasound : an Observational Transversal Study Conducted Using Images Registered From Patients (AIJV-I)
Acronym: AIJV-I
Status: Active, not recruiting | Type: Observational
Sponsor: Maggiore Bellaria Hospital, Bologna (Other)
Responsible Party: Principal Investigator, Nicola Parenti, MD, Maggiore Bellaria Hospital, Bologna
Other Study IDs: 725-2023-OSS-AUSLBObis
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hypervolemia; Hypovolemia
Keywords: reliability; internal jugular vein; ultrasound
MeSH Terms: conditions — Edema; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to test the inter-rater reliability among a group of ultrasound measurements of internal jugular vein using a group of images, registered in several acoustic views of neck of patients admitted in Medicine Department.

The main questions it aims to answer is: are there differences in recording echographic measurements of the internal jugular vein between different sonographers ?

DETAILED DESCRIPTION:
Dear Mrs/s, We intend to carry out medical scientific research in this Centre. It is a study of observation.. This study aims to measure the reliability (variability in recording measurements between two or more operators) of a new method, the ultrasound of a vein in the neck, called the internal jugular vein. This method could be used to better assess congestion (accumulation of fluid in the lung or tissues: vessels and skin) or lack of fluid in the veins, both possible causes of hospitalization.

We are proposing to you to participate in this study because you are hospitalized in the ward and this method allows to understand, together with other elements, the state of "volemia" (the amount of liquids present in your veins).

We decided to carry out this study because we would like to verify if the ultrasound of the internal jugular vein is reliable, that is it can be used by several operators without variations in the measurements . This would allow, after further studies, to use it in clinical practice for the management of people who may need fluid infusion or therapies to increase fluid removal.

The study aims to evaluate the reliability (variability in recording measurements between two or more operators) of ultrasound of a vein of the neck, called internal jugular vein In particular we would like to understand if there is a variability in the execution of the ultrasound of the jugular vein between several operators- doctors simultaneously to the same patient. In fact, this method is not currently used in current clinical practice, but if we demonstrate that it is reliable (ie more operators record the same measurements on the same patient , without variations), after further confirmation studies have been conducted , could be used in clinical practice. Its use could, in our view, improve the management of many situations, as it would allow doctors to understand whether the person examined is suffering from "congestion", that is, accumulation of water in the lungs and tissues or lack of fluids. This would allow the doctor to take appropriate therapies to reduce congestion or increase fluid.

During the hospitalization, on one occasion, will be submitted to an ultrasound examination of the neck on the right , simultaneously by two or three operators (doctors) . Each operator's examination should take about 10-15 minutes. So the time you spend on it should be 20-30 minutes. The examination will be carried out in bed, in his room with the back tilted 45 degrees and the neck slightly turned to the left.

The necessary treatment and examinations will be carried out and the reason for his admission will be continued.

There is no health risk, as ultrasound is a non-invasive examination based on ultrasound. The only discomfort is to be subjected for about thirty minutes to two or three consecutive examinations. There are no direct benefits to the participants. The study is oriented towards acquiring more scientific knowledge.

ELIGIBILITY:
Inclusion Criteria:

* patients, admitted to the Medicine Department of Hospital Maggiore in Bologna and eight expert sonographers

Exclusion Criteria:

* impossibility in providing consent, presence of central venous catheter in the internal jugular vein, thrombosis of the vein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include 2 populations:
  Patients admitted , for any causes, to the Medicine Department (we will record a group of 6 images that will be used by the sonographers).
  Sonographers from Medicine Department
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-09-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability of Internal Jugular Vein Ultrasound measures | From enrollment to the end of recording (within 2 months of starting the study)
  We will measure the variability in recording, among 8 sonographers, of 4 Ultrasound measures of Internal Jugular Vein : the antero-posterior diameters, the area, the aspect ratio and the collapsibility index

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Parenti, MD, Principal Investigator — Medicina Interna Hospital Maggiore Bologna
Locations (1):
- Hospital Maggiore, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Yes
I will share the study protocol.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: The criteria that must be met in order for data to be shared are:
  Clinical Researchers who conduct independent research Analyses on diagnostic accuracy of ultrasound methods Statistical methods for those analyses must be not approved by independent review.
  A proposal that describes planned analyses must be submitted and a data sharing agreement must be signed.
  Those documents can be submitted by sending a mail to nicola.parenti@ausl.bologna.it
URL: https://docs.google.com/document/d/10aop9iAeTrVKNpiofbG017R3AYAlCfFHVa0HPs6Y-00/edit?usp=sharing

REFERENCES:
- See also: Thelink of the Hospital of PI — https://www.ausl.bologna.it/
- Available data/document: Study Protocol — https://www.ausl.bologna.it/ — To send a request by mail